CLINICAL TRIAL: NCT04707079
Title: A Phase 2, Single Arm, Open Label, Multi-center Clinical Study of Dual PI3K-δ,γ Inhibitor Duvelisib in Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: A Safety and Efficacy Study of Duvelisib in Relapsed/Refractory Follicular Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE1801201901/PRO
Record Dates: First submitted 2020-04-24; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — duvelisib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Duvelisib (Experimental): Eligible subjects will be given duvelisib (15mg, 25mg), orally at a dose of 25 mg BID during each 28-day treatment cycle, for up to 12 cycles.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Eligible subjects will be given duvelisib orally at a dose of 25 mg BID during each 28-day treatment cycle, for up to 12 cycles.
  Other Names: COPIKTRA

SUMMARY:
This is a phase 2 clinical trial to evaluate the safety and efficacy of duvelisib as a monotherapy in subjects diagnosed with follicular lymphoma (FL) that is relapsed or refractory to either chemotherapy or radioimmunotherapy (RIT).

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-center clinical trial to evaluate the efficacy and safety of duvelisib administered to subjects who have been diagnosed with follicular lymphoma that is relapsed or refractory to either chemotherapy or RIT.

Subjects (n=57) will receive 25 mg duvelisib twice daily (BID) over the course of 28-day treatment cycles for up to 12 cycles.

After completing 12 treatment cycles of duvelisib, subjects may continue to receive additional cycles of duvelisib until disease progression or unacceptable toxicity. However, to receive additional cycles of duvelisib beyond 12 cycles, subjects must have evidence of response (CR, PR or SD) by the end of Cycle 12.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been fully informed and signed informed consent form.
2. Subjects must be adults (>/=18 years), male or female.
3. Subjects who have been defined as FL by histologic or cytologic diagnosis, and must have relapsed or been refractory (at least two prior regimens for FL).
4. Measurable disease with a lymph node or tumor mass ≥1.5 cm in at least one dimension by CT, PET/CT or MRI according to Lugano 2014 criteria.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Adequate renal and hepatic function.
7. Women of childbearing potential must have a negative serum or urine β human chorionic gonadotropin (βhCG) pregnancy test.
8. Willingness of male and female subjects who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study, including 30 days after the last dose of duvelisib.

Exclusion Criteria:

1. Grade 3B FL and/or clinical evidence of transformation to a more aggressive subtype of lymphoma.
2. Known hypersensitivity to the study drug duvelisib or excipients.
3. Previous treatment with a PI3K inhibitor or BTK inhibitor.
4. Prior history of allogeneic hematopoietic stem cell transplant (HSCT).
5. Prior chemotherapy, cancer immunosuppressive therapy, radiotherapy or other investigational agents within 4 weeks before the first dose of study drug.
6. Symptomatic central nervous system (CNS) Lymphoma.
7. Ongoing systemic bacterial, fungal, or viral infections at the time of initiation of study treatment.
8. Human immunodeficiency virus (HIV) infection.
9. Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection.
10. Hepatitis B or hepatitis C Infection.
11. History of stroke, unstable angina, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to first dose of study drug.
12. Female subjects who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR), | Within 7 days prior to initiating the next cycle of study treatment (i.e. Day -7 to Day 1) of Cycles 3, 5, 7, 9 (each cycle is 28 days) and at every fourth cycle thereafter (Cycle 13, 17, 21, etc.) up to the end of treatment, an average of 8 months.
  Defined as the best response of complete response/remission (CR) or partial response/remission (PR), according to the Cheson 2007 Criteria by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
ORR assessed by study sites according to the Cheson 2007 Criteria; | Within 7 days prior to initiating the next cycle of study treatment (i.e. Day -7 to Day 1) of Cycles 3, 5, 7, 9 (each cycle is 28 days) and at every fourth cycle thereafter (Cycle 13, 17, 21, etc.) up to the end of treatment, an average of 8 months.
ORR assessed respectively by study sites and IRC, according to the Lugano 2014 Criteria; | Within 7 days prior to initiating the next cycle of study treatment (i.e. Day -7 to Day 1) of Cycles 3, 5, 7, 9 (each cycle is 28 days) and at every fourth cycle thereafter (Cycle 13, 17, 21, etc.) up to the end of treatment, an average of 8 months.
Treatment-emergent adverse events (TEAEs), ECG measures, and changes in safety laboratory values; | Every 2-8 weeks; up to 30 days after the last dose of duvelisib.
Duration of Response; | Within 7 days prior to initiating the next cycle of study treatment (i.e. Day -7 to Day 1) of Cycles 3, 5, 7, 9 (each cycle is 28 days) and at every fourth cycle thereafter (Cycle 13, 17, 21, etc.) up to the end of treatment, an average of 8 months.
Progression-free survival; | Every 12 weeks; for an average response / progression follow-up of 2 years.
Overall survival; | Every 3 months; for an average survival follow-up of 3 years.
Time to response; | From the date of the first dose until the date of first documented complete response or partial response, assessed up to 2 years.
Maximum Plasma Concentration (ng/ml) for duvelisib and its metabolite IPI-656; | Every 4 weeks for 12 weeks.
Area under the Curve (ng*h/ml) for duvelisib and its metabolite IPI-656; | Every 4 weeks for 12 weeks
Elimination half life (h) for duvelisib and its metabolite IPI-656; | Every 4 weeks for 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China